CLINICAL TRIAL: NCT01087463
Title: Composite Nailing System for the Intramedullary Fixation of Humerus Fractures Without Intramedullary Reaming
Brief Title: Intramedullary Fixation of Humerus Fractures Without Intramedullary Reaming
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: N.M.B. Medical Applications Ltd (Industry)
Responsible Party: Gili Laufer, Hilel Yafe Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N.M.B. P_HY Q REV I 09.09
Record Dates: First submitted 2010-03-14; First posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-02

CONDITIONS: Humeral Fractures; Pathological Fractures
MeSH Terms: conditions — Humeral Fractures; Fractures, Spontaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (Experimental): In this single arm study, the Quantum nailing system will be used in all patients.
  Interventions: Device: Quantum

INTERVENTIONS:
Device: Quantum — Treatment of humerus fracture (according to the mentioned indications) with the Quantum Intramedullary Nailing System.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the composite Nail - the Quantum interlocking intramedullary nailing system in the reduction of humeral fractures.

DETAILED DESCRIPTION:
The study will include 20 patients who have an acute mid shaft diaphyseal humeral fracture due to injury. The patients will undergo lateral and AP X- ray evaluation of the fracture. Following General anesthesia, closed reduction of the fracture will be performed. It will be followed by nail insertion, percutaneously, according to standard surgical techniques, with the help of the insertion handle and without preliminary reaming. Following insertion the nail will be locked both distally and proximally using interlocking screws. The nail and screws insertion will be monitored by fluoroscopy. Patients will remain under follow up for 6 months following the procedure. In the follow up sessions the fracture will be evaluated by fluoroscopy or X-ray for correct bone alignment, callus formation, and fracture union.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old.
* Mid shaft diaphyseal fracture
* Acute fracture

Exclusion Criteria:

* Patients with metabolic or hormonal diseases that could affect bone healing such as diabetes.
* Ongoing infection in fracture site.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Bone union and callus formation,bone alignment, nail and screws resistance over time | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gili Laufer, Orthopedic, Principal Investigator — Hilel Yafe Medical Center
Locations (1):
- Hilel Yafe Medical Center, Hadera, Israel